CLINICAL TRIAL: NCT06346509
Title: A Phase 1, First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose and Food Effect Study of PORT-77 Administered Orally to Healthy Adult Participants
Brief Title: Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of PORT-77 Administered to Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Portal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PORT-77-101
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adult Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PORT-77 (Experimental): Healthy adult participants in each cohort will receive a single oral dose of PORT 77 or matching placebo on Day 1.
  Interventions: Drug: PORT-77
- Placebo (Placebo Comparator): Healthy adult participants in each cohort will receive a single oral dose of PORT 77 or matching placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PORT-77 — Healthy adult participants will receive a single oral dose of PORT 77.
  Arms: PORT-77
Drug: Placebo — Healthy adult participants will receive matching placebo on Day 1.
  Arms: Placebo

SUMMARY:
A First-in-Human 2-part, randomized, double-blind, placebo-controlled, single ascending dose, multiple ascending dose, and food effect, investigation of the administration of PORT-77 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* All healthy adult participants must be willing and able to follow protocol-specified assessments.
* Healthy based on no clinically significant medical history, physical examination, laboratory profiles, vital signs, and Electrocardiograms (ECGs), as deemed by the Principal Investigator (PI) or designee.

Exclusion Criteria:-

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* Female subject with a positive pregnancy test at the screening visit or at first check-in or who is lactating.
* Participation in another clinical study within 60 days or within 10 half-lives (if known), prior to the first dosing, whichever is longer, or previous participation in another PORT 77 study or study part.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Number of incidence and severity of adverse events (AEs) as a measure of safety and tolerability of PORT-77 (Part I) | Day 8
Number of incidence and severity of AEs as a measure of safety and tolerability of PORT-77 (Part II) | Day 21

SECONDARY OUTCOMES:
Plasma concentration of a single-dose of PORT-77 (Part I) | Day 8
Plasma concentration of the steady-state of PORT-77 (Part II) | Day 21
Plasma concentration of PORT-77 by effect of a standardized high-fat/high-calorie meal (Part I) | Day 4
Evaluate effects of single doses of PORT-77 on ECG parameters (Part I) | Day 8
Evaluate effects of single doses of PORT-77 on ECG parameters (Part II) | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Portal Therapeutics, Chief Medical Officer, Study Director — Portal Therapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No